CLINICAL TRIAL: NCT06764589
Title: Liquid Micro-biopsy: a Novel Approach to Study Tumor Microenvironment From the Peripheral Blood
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO-biopsy
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Acute Myelocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Periferal blood, Bone marrow aspirate and bone marrow biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective multicentre, tissue-based, non-profit study that includes two enrolling centres: Operating Unit (OU) No. 1 of Haematology and OU No. 2 of Medical Oncology, both at the IRCCS Azienda Ospedaliera-Universitaria di Bologna (AOUBO). Given the rarity of the pathology investigated and the lack of evidence from the literature, the study should be considered exploratory, aimed at providing provisional evidence and generating hypotheses that could be tested in future studies.

The study involves the collection of peripheral blood samples from healthy volunteers (HD) matched for sex/age (n=30; Group 1) and patients with acute myeloid leukaemia at diagnosis (n=30; Group 2) at UO1 and patients with visceral sarcoma with measurable disease (n=30; Group 3) at UO2.

Specifically, peripheral blood (equal to 60 mL) from healthy volunteers will be collected after obtaining the signed informed consent of the volunteers of the Associazione Onlus AIL Bologna ODV.

From all participants in Groups 2 and 3, 60 mL of peripheral blood and 20 mL of bone marrow blood will be collected at routine clinical examinations. Bone biopsies (10 sections) will also be collected from Group 2 patients. All samples will be collected at the time of diagnosis (T0). All samples will be centralised at the Haematology Unit, IRCCS AOUBO and submitted for laboratory analysis.

For patients with acute myeloid leukaemia, responses to treatment will be assessed on the basis of standard criteria according to the recommendations of the European LeukemiaNet of 2022 (Döhner H et al, Blood 2022). Clinical response for sarcoma patients according to the international RECIST imaging criteria assessed by routine computed tomography or magnetic resonance imaging scans.

DETAILED DESCRIPTION:
Survival of AML is globally poor, with an overall survival at 5 years largely inferior to 50%. The diagnosis of several diseases, such as AML relies on invasive procedures. An increasing amount of evidence supports the straightforward relations between bone marrow (BM) biopsies and blood in hematological malignancies, including AML. Novel approaches to the characterization of TME have been developed. In this regard, scRNA-seq analysis emerged as a potent tool, capable of profoundly characterizing genomic profiles at the single-cell level. However, ST have the potential to improve our understanding of TME composition and cellular interactions, representing a powerful tool capable of identifying cell types and gene expression profiles on a structural and spatial level.

Since the question of a comprehensive characterization of tumor heterogeneity and cell-cell interactions is still unsolved, new ways to detect its modulation using blood are highly warranted for tumor diagnosing and monitoring. Indeed, conventional and invasive methods are insufficient to decipher the heterogeneous nature of tumors. Based on these premises, the driving hypothesis of the study is that performing an in-parallel analysis on both circulating cells and EVs might provide a broader characterization of the genomic landscape of tumors than using cells themselves. The integration of LB within the clinical management of cancer patients may represent an essential step towards a deeper understanding of cancer biology. It might have important implications for better disease monitoring and improved drug development.

ELIGIBILITY:
Inclusion Criteria:

* For HD:

  * Age ≥ 18 years
  * Volunteer in general good health, free from any disease or serious illness
  * Signed written informed consent to study participation and personal data processing

For AML patients:

* Age ≥ 18 years
* New diagnosis of AML according to World Health Organization 2022 criteria
* Front-line treatment according to routine clinical practice
* Signed written informed consent to study participation and personal data processing

For sarcoma patients:

* Age ≥ 18 years
* Diagnosis of visceral soft tissue sarcoma according to World Health Organization 2021 criteria in metastatic setting
* Signed written informed consent to study participation and personal data processing

Exclusion Criteria:

* For HD:

  * None

For AML and sarcoma patients:

* Acute promyelocytic leukemia (for AML)
* Known AML with central nervous system involvement (for AML)
* Visceral sarcoma in adjuvant setting (for sarcoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The planned population size for the study is 90 prospectively enrolled patients, 30 for each of the three study groups. No sample size calculations were performed due to the exploratory nature of this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
1. Malignant signals (cell subsets and EV markers) | At diagnosis (T0)
  The percentages of positive/negative cells for each marker and the markers' geometric means are measured by flow cytometry and defined by negative control or by the value detected by HD (group 1) versus AML or sarcoma patients (group 2-3).

SECONDARY OUTCOMES:
2. Transcriptomic profile in cells and EVs | At diagnosis (T0)
  Gene count and transcript quantifications and computational analyses (deconvolution) are collected in HD (group 1) and AML or sarcoma patients (group 2-3).

OTHER OUTCOMES:
3. Tissue characterization and spatial profiling | At diagnosis (T0)
  Marker expression in tumoral cells are recorded as the percentage (%) of positive cells in relation to the overall neoplastic population by conventional immunohistochemistry and morphological analysis.
  Gene and proteomic expression for specific microenvironmental markers are processed by imaging and scored as the mean number of positive cells/mm2.
4. Clinical response prediction for AML and sarcoma patients from LB or spatial data | At diagnosis (T0) At the first response evaluation after therapy, according to routine clinical practice
  For AML patients, clinical responses are assessed as follows:
  * Complete Remission (CR): BM blasts <5%; absence of circulating blasts or blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count ≥1.0 x 109/L (1,000/μL); platelet count ≥100 x 109/L (100,000/μL)
  * CR with partial hematologic recovery (CRh): absolute neutrophil count ≥0.5 x 109/L (500/μL) and platelet count ≥50 x 109/L (50,000/μL), otherwise all other CR criteria met
  * CR with incomplete hematologic recovery (CRi): All CR criteria except for residual neutropenia <1.0 x 109/L (1,000/μL) or thrombocytopenia <100 x 109/L (100,000/μL)
  * Refractoriness: No CR, CRh or CRi For sarcoma patients, clinical responses are assessed according to international imaging RECIST criteria evaluated by routine computed tomography or magnetic resonance imaging scans.
  Prediction of clinical response at the diagnosis are elaborated by computational method and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - IRCCS Azienda-Ospedaliero Universitaria di Bologna, Bologna